CLINICAL TRIAL: NCT01329393
Title: Benefits Management for People With Psychiatric Disabilities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0910005874; R34MH083894 (NIH)
Record Dates: First submitted 2011-02-02; First posted 2011-04-05 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2014-07

CONDITIONS: Dual Diagnosis; Schizophrenia; Bipolar Disorder
Keywords: Disability; Social Security; Representative Payee
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benefits Management (Experimental): Money-management intervention consisting of brief advice on budgeting, assessment of ability to follow a budget, and assessment of need for a representative payee.
  Interventions: Behavioral: Benefits Management
- Illness Management and Recovery (Active Comparator)
  Interventions: Behavioral: Illness Management and Recovery

INTERVENTIONS:
Behavioral: Benefits Management — Money-management intervention consisting of brief advice on budgeting, assessment of ability to follow a budget, and assessment of need for a representative payee.
  Arms: Benefits Management
Behavioral: Illness Management and Recovery — Recovery Oriented Training in Biopsychosocial Model of Stress and How to Cope with Stress
  Arms: Illness Management and Recovery

SUMMARY:
This stage 1 clinical trial will determine pilot efficacy, develop a therapy manual, and collect qualitative data concerning a brief money management intervention for people disabled by psychiatric illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Has received treatment for a psychiatric disorder within 60 days of enrollment
* Receives SSI or SSDI payments totaling at least $600 per month
* Has an identified outpatient clinician
* Either i) Homeless within the past 3 months. Homeless is defined as having spent at least seven days in a shelter, outdoors (e.g. in a park, in a car), in a public or abandoned building (e.g. train station), or temporarily (less than a continuous month) housed by family or friends OR ii) Hospitalized within the past 3 months

Justification for Inclusion Criteria: Homelessness and hospitalization are common reasons for payee assignment (Conrad, Matters et al. 1998). In a prior study, we found that a high proportion of hospitalized inpatients meet criteria for needing a payee (Rosen, Rosenheck et al. 2002a). There is no point enrolling clinically stable outpatients in this study because they are unlikely to need payees.

Exclusion Criteria:

* Already has a conservator or representative payee
* An application to assign a payee or conservator has been initiated
* Unable to speak and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in the Summed score on the Heinrich-Carpenter Quality of Life Measure | Change from Week 0 to Week 24
  The Heinrich-Carpenter Quality of Life score is derived by summing ratings of individual items after a semi-structured interview. The possible score on any given interview is 0-126. It is a global measure of social functioning with higher scores indicating better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Marc I. Rosen, M.D., Principal Investigator — Yale University
Locations (1):
- Institute of Living, Hartford, Connecticut, United States